CLINICAL TRIAL: NCT01986101
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study of SM-13496 for the Treatment of Bipolar I Depression.
Brief Title: A Phase III Study of SM-13496 in Patients With Bipolar I Depression.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1002001; JapicCTI-132318 (Registry Identifier: JAPIC Clinical Trials Information); 2013-003038-34 (EudraCT Number)
Record Dates: First submitted 2013-11-04; First posted 2013-11-18 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): once daily orally
  Interventions: Drug: Placebo
- SM-13496 20 - 60 mg/day (Experimental): once daily orally
  Interventions: Drug: SM-13496
- SM-13496 80 - 120 mg/day (Experimental): once daily orally
  Interventions: Drug: SM-13496

INTERVENTIONS:
Drug: Placebo — Placebo comparator
  Arms: Placebo
Drug: SM-13496 — SM-13496 20mg for Days 1-7 and beginning Day 8 flexibly dosed 20-60 mg/day for Weeks 2-6
  Other Names: Lurasidone HCl
  Arms: SM-13496 20 - 60 mg/day
Drug: SM-13496 — SM-13496 20 mg/day for Days 1-2, 40 mg/day for Days 3-4, 60 mg/day for Days 5-6, 80 mg/day on Day 7 and beginning Day 8 flexibly dosed 80-120 mg/day for Weeks 2-6
  Other Names: Lurasidone HCl
  Arms: SM-13496 80 - 120 mg/day

SUMMARY:
The study evaluates the efficacy and safety of SM-13496 compared with placebo in patients with Bipolar I Depression.

DETAILED DESCRIPTION:
The primary objective is to compare the efficacy of SM-13496 (20-60 or 80-120 mg/day) monotherapy with that of placebo in patients with depressive symptoms associated with bipolar I disorder by assessing the change from baseline in the MADRS total score at Week 6.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were fully informed of and understand the objectives, procedures, and possible benefits and risks of the study and who provided written voluntary consent to participate in the study.
* Outpatients aged 18 through 74 years at the time of consent
* Patients meets DSM-IV-TR criteria for bipolar I disorder, most recent episode depressed (≥ 4 weeks and less than 12 months) without psychotic features.

Exclusion Criteria:

* Patients with imminent risk of suicide or injury to self, others, or property.
* Patients who had been hospitalized because of a manic or mixed episode within 60 days prior to screening.
* Patients who are otherwise considered ineligible for the study by the investigator.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Drug Development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (8):
- Japan 76 sites, Tokyo, Japan
- Lithuania 3 sites, Kaunas, Lithuania
- Malaysia 5 sites, Kuala Lumpur, Malaysia
- Philippines 4 sites, Manila, Philippines
- Russia 19 sites, Moscow, Russia
- Slovakia 5 sites, Žilina, Slovakia
- Taiwan 7 sites, Taipei, Taiwan
- Ukraine 9 sites, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kato T, Ishigooka J, Miyajima M, Watabe K, Fujimori T, Masuda T, Higuchi T, Vieta E. Double-blind, placebo-controlled study of lurasidone monotherapy for the treatment of bipolar I depression. Psychiatry Clin Neurosci. 2020 Dec;74(12):635-644. doi: 10.1111/pcn.13137. Epub 2020 Sep 24. PMID 32827348
- [Derived] Hopkins SC, Tomioka S, Szabo ST, Koblan KS. A clinical trial inclusion criteria to enrich for patients presenting with canonical symptom structure in bipolar depression. Contemp Clin Trials. 2024 Oct;145:107644. doi: 10.1016/j.cct.2024.107644. Epub 2024 Aug 3. PMID 39098761
- [Derived] Kishi T, Nakamura H, Kato T, Iwata N. A diagnostic test to examine early improvement as a predictor of later response to lurasidone in bipolar depression. Neuropsychopharmacol Rep. 2023 Mar;43(1):137-140. doi: 10.1002/npr2.12319. Epub 2023 Jan 12. PMID 36632763
- [Derived] Kishi T, Yoshimura R, Sakuma K, Okuya M, Iwata N. Lurasidone, olanzapine, and quetiapine extended-release for bipolar depression: A systematic review and network meta-analysis of phase 3 trials in Japan. Neuropsychopharmacol Rep. 2020 Dec;40(4):417-422. doi: 10.1002/npr2.12137. Epub 2020 Sep 9. PMID 32902200

RESULTS

PARTICIPANT FLOW:
Groups:
- SM-13496 20 - 60 mg/Day: once daily orally
  SM-13496: SM-13496 20mg for Days 1-7 and beginning Day 8 flexibly dosed 20-60mg/day for Weeks 2-6
Period: Overall Study
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day
Started | 172 | 184 | 169
Intent-to-Treat Population | 171 | 182 | 169
Safety Population | 172 | 184 | 169
Completed | 139 | 157 | 137
Not Completed | 33 | 27 | 32

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population is analyzed.
Groups:
- Placebo: once daily orally
  Placebo
- SM-13496 20 - 60 mg/Day: once daily orally
  SM-13496 (lurasidone HCl): SM-13496 20 mg/day for Days 1-7 and beginning Day 8 flexibly dosed 20-60 mg/day for Weeks 2-6
- SM-13496 80 - 120 mg/Day: once daily orally
  SM-13496 (lurasidone HCl): SM-13496 20 mg/day for Days 1-2, 40 mg/day for Days 3-4, 60 mg/day for Days 5-6, 80 mg/day on Day 7 and beginning Day 8 flexibly dosed 80-120 mg/day for Weeks 2-6
- Total: Total of all reporting groups
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day | Total
Number analyzed (Participants) | 171 | 182 | 169 | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.64) | 42.6 (12.86) | 43.2 (12.78) | 42.4 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 95 | 88 | 277
  Male | 77 | 87 | 81 | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 94 | 105 | 103 | 302
  Asian | 77 | 77 | 66 | 220
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 60 | 65 | 53 | 178
  Philippines | 5 | 3 | 3 | 11
  Taiwan | 5 | 3 | 4 | 12
  Ukraine | 43 | 43 | 45 | 131
  Malaysia | 7 | 6 | 6 | 19
  Slovakia | 5 | 7 | 4 | 16
  Lithuania | 2 | 4 | 4 | 10
  Russia | 44 | 51 | 50 | 145
Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — Montogomery-Asberg Depression Rating Scale (MADRS) is a clinician-rated assessment of a subject's level of depression. The MADRS total score ranges from a minimum of 0 to a maximum of 60. Low scores indicate a better outcome and high scores indicate a worse outcome. The MADRS total score contains 10 items. The total score is computed as the sum of the scores for the 10 items.
  units on a scale | 30.9 (5.39) | 30.6 (5.57) | 30.8 (5.09) | 30.8 (5.35)
Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) Score (Depression) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) score (depression) is a clinician-rated assessment of a subject's level of depression. The score ranges from a minimum of 1 to a maximum of 7. Low scores indicate a better outcome and high scores indicate a worse outcome.
  units on a scale | 4.60 (0.690) | 4.57 (0.700) | 4.58 (0.603) | 4.58 (0.666)
Sheehan Disability Scale (SDS) total score [Mean (Standard Deviation); unit: units on a scale] — Sheehan Disability Scale (SDS) total score is a subject-rated assessment of a subject's level of functional impairment in work/school, social life and family life/home responsibilities.
  The SDS total score ranges from a minimum of 0 to a maximum of 30. Low scores indicate a better outcome and high scores indicate a worse outcome. The SDS total score contains 3 items. The total score is computed as the sum of the scores for the 3 items. Population: SDS total score was evaluated in most subjects.
  units on a scale
    number analyzed (Participants) | 141 | 154 | 127 | 422
    (all) | 19.9 (5.22) | 19.4 (5.29) | 19.8 (5.58) | 19.7 (5.35)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 6
Description: Montgomery-Asberg Depression Rating Scale (MADRS)is a clinician-rated assessment of a subject's level of depression.
  The MADRS total score ranges from a minimum of 0 to a maximum of 60. For the MADRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The MADRS contains ten (10) items. The total score is computed as the sum of the scores for the 10 items.
Time Frame: Baseline to 6 weeks
Population: Intention-to-treat population is analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- SM-13496 20 - 60 mg/Day: once daily orally
  SM-13496: SM-13496 20 mg/day for Days 1-7 and beginning Day 8 flexibly dosed 20-60 mg/day for Weeks 2-6
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day
Number analyzed (Participants) | 171 | 182 | 169
units on a scale | -10.6 (0.72) | -13.6 (0.69) | -12.6 (0.73)
Statistical Analysis 1: Comparison: Placebo vs SM-13496 20 - 60 mg/Day; Test type: Superiority; p = 0.007, Mixed Models Analysis — Hochberg-adjusted; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-4.9 to -1.0], Standard Error of Mean 1.00 — A negative difference in least square mean change from baseline between SM-13496 group and placebo indicates a greater improvement in the SM-13496 group over the placebo group
Statistical Analysis 2: Comparison: Placebo vs SM-13496 80 - 120 mg/Day; Test type: Superiority; p = 0.057, Mixed Models Analysis — Hochberg-adjusted; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.0 to 0.1], Standard Error of Mean 1.03 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in the CGI-BP-S (Depression) Score at Week 6
Description: Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) score (depression) is a clinician-rated assessment of a subject's level of depression.
  The CGI depression score ranges from a minimum of 1 to a maximum of 7. For the CGI depression score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
Time Frame: Baseline to 6 weeks
Population: Intention-to-treat population is analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day
Number analyzed (Participants) | 171 | 182 | 169
units on a scale | -1.11 (0.092) | -1.51 (0.088) | -1.41 (0.093)
Statistical Analysis 1: Comparison: Placebo vs SM-13496 20 - 60 mg/Day; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.65 to -0.15], Standard Error of Mean 0.127 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SM-13496 80 - 120 mg/Day; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.56 to -0.05], Standard Error of Mean 0.130 — A negative difference in least square mean change from baseline between SM-13496 group and placebo indicates a greater improvement in SM-13496 group over the placebo group

3. Secondary Outcome: Change From Baseline in the SDS Total Score at Week 6 (LOCF)
Description: Sheehan Disability Scale (SDS) total score is a subject-rated assessment of a subject's level of functional impairment in work/school, social life and family life/home responsibilities.
  The SDS total score ranges from a minimum of 0 to a maximum of 30. For the SDS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The SDS contains three (3) items. The total score is computed as the sum of the scores for the 3 items.
Time Frame: Baseline to 6 weeks
Population: Intention-to-Treat Population is analyzed. Values were missing for some subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day
Number analyzed (Participants) | 128 | 147 | 124
units on a scale | -5.7 (0.66) | -7.6 (0.62) | -6.8 (0.67)
Statistical Analysis 1: Comparison: Placebo vs SM-13496 20 - 60 mg/Day; Test type: Superiority; p = 0.037, ANCOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.6 to -0.1], Standard Error of Mean 0.89 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SM-13496 80 - 120 mg/Day; Test type: Superiority; p = 0.223, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.9 to 0.7], Standard Error of Mean 0.92 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in the YMRS Total Score at Week 6
Description: YMRS (Young Mania Rating Scale) is a clinician-rated assessment of the severity of mania in subjects with a diagnosis of bipolar disorder.
  The YMRS total score ranges from a minimum of 0 to a maximum of 60. For the YMRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The YMRS contains eleven (11) items. The total score is computed as the sum of the scores for the 11 items.
Time Frame: Baseline to 6 weeks
Population: Intention-to-Treat Population is analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day
Number analyzed (Participants) | 171 | 182 | 169
units on a scale | -0.51 (0.190) | -0.98 (0.180) | -0.99 (0.191)
Statistical Analysis 1: Comparison: Placebo vs SM-13496 20 - 60 mg/Day; Test type: Superiority; p = 0.076, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.98 to 0.05], Standard Error of Mean 0.262 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SM-13496 80 - 120 mg/Day; Test type: Superiority; p = 0.075, Mixed Models Analysis; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.01 to 0.05], Standard Error of Mean 0.269 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in the HAM-A Total Score at Week 6 (LOCF)
Description: The Hamilton Rating Scale for Anxiety (HAM-A) scale is a rating scale developed to quantify the severity of anxiety symptomatology.
  The HAM-A total score ranges from a minimum of 0 to a maximum of 56. For the HAM-A total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The HAM-A contains fourteen (14) items. The total score is computed as the sum of the scores for the 14 items.
Time Frame: Baseline to 6 weeks
Population: Intention-to-treat population is analyzed. Values were missing for some subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day
Number analyzed (Participants) | 164 | 179 | 167
units on a scale | -5.7 (0.51) | -7.4 (0.49) | -6.4 (0.50)
Statistical Analysis 1: Comparison: Placebo vs SM-13496 20 - 60 mg/Day; Test type: Superiority; p = 0.016, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.1 to -0.3], Standard Error of Mean 0.70 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SM-13496 80 - 120 mg/Day; Test type: Superiority; p = 0.294, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.1 to 0.7], Standard Error of Mean 0.71 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Safety population is analyzed.
Arm/Group | Placebo | SM-13496 20 - 60 mg/Day | SM-13496 80 - 120 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/184 | 0/169
Serious Adverse Events (participants affected / at risk) | 5/172 | 2/184 | 4/169
Other Adverse Events (participants affected / at risk) | 44/172 | 49/184 | 75/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=172) | SM-13496 20 - 60 mg/Day (N=184) | SM-13496 80 - 120 mg/Day (N=169)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=172) | SM-13496 20 - 60 mg/Day (N=184) | SM-13496 80 - 120 mg/Day (N=169)
Nausea (Gastrointestinal disorders) | 10 (13) | 12 (13) | 20 (23)
Nasopharyngitis (Infections and infestations) | 8 (8) | 10 (10) | 6 (6)
Akathisia (Nervous system disorders) | 11 (12) | 24 (27) | 40 (46)
Headache (Nervous system disorders) | 15 (22) | 5 (7) | 9 (11)
Parkinsonism (Nervous system disorders) | 4 (7) | 4 (4) | 10 (19)
Somnolence (Nervous system disorders) | 7 (8) | 7 (7) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT01986101/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT01986101/SAP_001.pdf